CLINICAL TRIAL: NCT02333539
Title: Adherence Intervention to Promote Optimal Use of Insulin Pumps in Adolescents
Brief Title: Adherence Intervention to Promote Optimal Use of Insulin Pumps in Adolescents With Type 1 Diabetes
Acronym: Pump It Up!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0965
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored feedback (Experimental): Participants are provided a Tailored Feedback report based on data downloaded from their insulin pumps. Summaries are provided about insulin pump adherence behaviors and recommendations for improvement are made.
  Interventions: Behavioral: Adherence behaviors and recommendations for improvement.
- Problem Solving (Experimental): Participants receive a problem-solving session based on data downloaded from their insulin pumps. An insulin pump adherence behavior that needs improvement is targeted; goals are set and solutions generated.
  Interventions: Behavioral: Adherence behavior that needs improvement is targeted
- Treatment as Usual (No Intervention): Standard of care as provided by the endocrinologist occurs.

INTERVENTIONS:
Behavioral: Adherence behaviors and recommendations for improvement.
  Arms: Tailored feedback
Behavioral: Adherence behavior that needs improvement is targeted
  Arms: Problem Solving

SUMMARY:
The overall objective of this study is to address the critical need of improving insulin pump adherence in adolescents with Type 1 Diabetes (T1D) by providing personalized intervention using evidence-based techniques during routine diabetes clinic visits at point of care.

DETAILED DESCRIPTION:
To achieve optimal use of the insulin pump, patients must engage in frequent Blood Glucose Monitoring (BGM) and insulin bolusing, and have an understanding of their relationship. BGM must occur and then it must be followed by a decision about what to do (or not do) regarding insulin bolusing. If insulin bolusing occurs in the absence of BGM, hypoglycemia and less than ideal glycemic control can occur. Of the few insulin pump adherence studies, only very basic adherence behaviors such as BGM and insulin bolusing frequency or number of hypoglycemic events have been reported.

The overall objective of this study is to address the critical need of improving insulin pump adherence in adolescents with T1D by providing personalized intervention using evidence-based techniques during routine diabetes clinic visits at point of care.

ELIGIBILITY:
Inclusion Criteria:

* ages 10-17 years
* type 1 diabetes diagnosis at least 1 year
* use insulin pump

Exclusion Criteria:

* developmental delay

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Frequency of Insulin Pump Adherence Behaviors | every 3 months up to 12 months
  Frequency of blood glucose monitoring per day; frequency of carbohydrate inputs per day; frequency of insulin boluses per day; frequency of insulin boluses that follow a high (>150 mg/dL) or very high (>250mg/dL) blood glucose result.

SECONDARY OUTCOMES:
Change in Glycemic Control (A1C) | every 3 months up to 12 months
  Glycemic control (A1C) will be measured with a Siemens Healthcare Diagnostics DCA Vantage, which is National Glycohemoglobin Standardization Program certified as having documented traceability to the Diabetes Control and Complications Trial Reference Method; range 4.2-6.5%.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Driscoll, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- Florida State University, Tallahassee, Florida, United States